CLINICAL TRIAL: NCT01034969
Title: Icatibant Outcome Survey (IOS) Registry
Brief Title: Firazyr® Patient Registry (Icatibant Outcome Survey - IOS)
Status: Completed | Type: Observational
Sponsor: Shire (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: JE049-5134
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Hereditary Angioedema (HAE)
Keywords: Hereditary angioedema
MeSH Terms: conditions — Angioedemas, Hereditary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with hereditary angioedema (HAE): All participants with hereditary angioedema (HAE) who are administered Cinryze (C1 inhibitor [human]) or Firazyr (Icatibant) for the treatment or prevention of angioedema attacks in routine clinical practice will be included into the study.

SUMMARY:
The Icatibant Outcome Survey (IOS) is a prospective, observational disease registry designed to document the routine clinical outcomes over time in participants with angioedema treated with Firazyr® (icatibant) and/or Cinryze® (C1 inhibitor [human]) in countries where it is currently approved. The data collected will be used to evaluate the safety of Firazyr (icatibant) and Cinryze (C1 inhibitor [human]) in routine clinical practice and as a data source for post-marketing investigations.

DETAILED DESCRIPTION:
The Icatibant Outcome Survey (IOS) is a multicenter, prospective, observational study for participants treated with Firazyr (icatibant) and/or Cinryze (C1 inhibitor [human]) in countries where it is currently approved. The entry of participants in the Icatibant Outcome Survey (IOS) is at the discretion of the physician and the participant and is not a pre-requisite for prescribing Firazyr (icatibant) or Cinryze (C1 inhibitor [human]).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of at least 1 of the following:

   * Hereditary angioedema (HAE) type I or II
   * HAE with normal C1 inhibitor
   * ACE-I-induced angioedema
   * Non-histaminergic idiopathic angioedema
   * Acquired angioedema.
2. Signed and dated written informed consent from the participant or, for participants aged less than(<)18 years (or as per local regulation, such as <16 years in the United Kingdom [UK]), parent and/or participants legally authorized representative (LAR), and assent of the minor where applicable.
3. At sites only participating in the drug registry, participants must have taken at least 1 dose of Firazyr (Icatibant) or Cinryze (C1 inhibitor [human]).
4. Enrolled participants in Germany taking Firazyr (Icatibant) or Cinryze (C1 inhibitor [human]) will only use the respective product in accordance with the product label.

Exclusion Criteria:

1. Participants enrolled in clinical trials where the product is blinded or where the product under investigation is for the treatment of HAE, ACE-I-induced angioedema, non-histaminergic idiopathic angioedema, or acquired angioedema.
2. Participants enrolled in another Shire-sponsored registry involving products for the treatment of HAE, ACE-I-induced angioedema, non-histaminergic idiopathic angioedema, or acquired angioedema. An exception applies to participants enrolled in the Shire lanadelumab ENABLE study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with Type I or II HAE, and, where applicable, with angiotensin-converting enzyme inhibitor (ACE-I)-induced angioedema, non-histaminergic idiopathic angioedema, or acquired angioedema, irrespective of treatment and/or other treatments and also participants who have taken at least 1 dose of Firazyr (Icatibant) or Cinryze (C1 inhibitor [human]) will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1761 (Actual)
Dates: Start 2009-07-10 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Cardiac Ischemia Events in Participants Predisposed to Cardiac Ischemia Events With Concomitant Firazyr (Icatibant) Administration | From enrollment through study participation (Approximately 13 years)
  Incidence of cardiac ischemia events in participants predisposed to cardiac ischemia events with concomitant Firazyr (Icatibant) administration will be assessed.
Incidence of Hypotension for Firazyr (Icatibant) | From enrollment through study participation (Approximately 13 years)
  Incidence of hypotension for Firazyr (Icatibant) will be assessed.
Incidence of Swelling of Mucous Membranes for Firazyr (Icatibant) | From enrollment through study participation (Approximately 13 years)
  Incidence of swelling of mucous membranes for Firazyr (Icatibant) will be assessed.
Incidence of Bronchoconstriction for Firazyr (Icatibant) | From enrollment through study participation (Approximately 13 years)
  Incidence of bronchoconstriction for Firazyr (Icatibant) will be assessed.
Incidence of Aggravation of Pain for Firazyr (Icatibant) | From enrollment through study participation (Approximately 13 years)
  Incidence of aggravation of pain for Firazyr (Icatibant) will be assessed.
Sexual Hormones Level Measurements- Tanner Staging for Firazyr (Icatibant) | From enrollment through study participation (Approximately 13 years)
  Effects on sexual maturation in pubertal adolescents will be measured using Tanner staging (pubic hair stage and genital breast stage) for Firazyr (Icatibant).
Time to Complete Resolution of the Firazyr (Icatibant)-Treated Laryngeal Attacks | From enrollment through study participation (Approximately 13 years)
  Time to complete resolution of the laryngeal attacks will be assessed. It is defined as the time between the first injection of treatment and the complete resolution of all symptoms.
Incidence of Adverse Events (AE) Related to Firazyr (Icatibant)-Treated Laryngeal Attacks | From enrollment through study participation (Approximately 13 years)
  An AE is defined as any noxious, pathologic, or unintended change in anatomical, physiologic, or metabolic function as indicated by physical signs, symptoms, or laboratory changes occurring in the registry, whether or not considered product-related. This includes an exacerbation of a pre-existing condition.
Incidence of Adverse Drug Reactions (ADR) for Firazyr (Icatibant) | From enrollment through study participation (Approximately 13 years)
  An ADR is a response to a medicinal product that is noxious and unintended and that occurs at doses normally used in man for prophylaxis, diagnosis, and treatment of disease or for the restoration, correction, or modification of physiological function.
Incidence of Serious Adverse Events (SAE) for Firazyr (Icatibant) | From enrollment through study participation (Approximately 13 years)
  An AE or ADR that meets 1 or more of the following criteria or outcomes is classified as an SAE whether considered to be related to the pharmaceutical product or not: death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; a persistent or significant disability or incapacity; a congenital anomaly or birth defect; important medical events.
Incidence of Pregnancy and Lactation Events During Firazyr (Icatibant) Exposure | From enrollment through study participation (Approximately 13 years)
  The incidence of pregnancy or lactation events coinciding with exposure to Firazyr (Icatibant) will be summarized by angioedema treatment and subgroup.
Incidence of Adverse Events (AE) for Cinryze (C1 Inhibitor [Human]) | From enrollment through study participation (Approximately 13 years)
  An AE is defined as any noxious, pathologic, or unintended change in anatomical, physiologic, or metabolic function as indicated by physical signs, symptoms, or laboratory changes occurring in the registry, whether or not considered product-related. This includes an exacerbation of a pre-existing condition.
Incidence of Adverse Drug Reactions (ADR) for Cinryze (C1 Inhibitor [Human]) | From enrollment through study participation (Approximately 13 years)
  An ADR is a response to a medicinal product that is noxious and unintended and that occurs at doses normally used in man for prophylaxis, diagnosis, and treatment of disease or for the restoration, correction, or modification of physiological function.
Incidence of Serious Adverse Events (SAE) for Cinryze (C1 Inhibitor [Human]) | From enrollment through study participation (Approximately 13 years)
  An AE or ADR that meets 1 or more of the following criteria or outcomes is classified as an SAE whether considered to be related to the pharmaceutical product or not: death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; a persistent or significant disability or incapacity; a congenital anomaly or birth defect; important medical events.
Incidence of Thrombotic or Thromboembolic Events for Cinryze (C1 Inhibitor [Human]) | From enrollment through study participation (Approximately 13 years)
  Thrombotic or thromboembolic events will be reported as SAEs and will include, but are not limited to, established diagnoses of any of the following: renal allograft arterial or venous thrombosis; deep vein thrombosis; myocardial infarction; pulmonary embolism; Ischemic cerebrovascular accident (stroke)- cerebrovascular accident exclusive of cerebrovascular hemorrhage (subarachnoid or subdural hemorrhage); any large vessel thrombosis; thrombophlebitis; catheter-related thrombotic events (including clotted dialysis access grafts) will be assessed.
Incidence of Pregnancy and Lactation Events During Cinryze (C1 Inhibitor [Human]) Exposure | From enrollment through study participation (Approximately 13 years)
  The incidence of pregnancy or lactation events coinciding with exposure to Cinryze (C1 inhibitor [human]) will be summarized by angioedema treatment and subgroup.
Drug Exposure Data for Cinryze (C1 Inhibitor [Human]) | From enrollment through study participation (Approximately 13 years)
  Drug exposure data for Cinryze (C1 inhibitor [human]) for prophylaxis, pre-procedural, and acute treatments will be reported.
Frequency of Hereditary Angioedema (HAE) Attacks in Participants Treated With Cinryze (C1 Inhibitor [Human]) | From enrollment through study participation (Approximately 13 years)
  Frequency of HAE attacks in participants treated with Cinryze (C1 inhibitor [human]) will be assessed.
Severity of Hereditary Angioedema Attacks in Participants Treated With Cinryze (C1 Inhibitor [Human]) | From enrollment through study participation (Approximately 13 years)
  Severity of HAE attacks in participants treated with Cinryze (C1 inhibitor [human]) will be assessed.
Anatomic Location of Hereditary Angioedema Attacks in Participants Treated With Cinryze (C1 Inhibitor [Human]) | From enrollment through study participation (Approximately 13 years)
  Anatomic location of HAE attacks in participants treated with Cinryze (C1 inhibitor [human]) will be assessed.
Outcome of Severe or Laryngeal Hereditary Angioedema Attacks in Participants Treated With Cinryze (C1 Inhibitor [Human]) | From enrollment through study participation (Approximately 13 years)
  Outcome of severe or laryngeal HAE attacks in participants treated with Cinryze (C1 inhibitor [human]) will be assessed.
Outcome of Hereditary Angioedema Attacks for Treatment With Cinryze (C1 Inhibitor [Human]) | From enrollment through study participation (Approximately 13 years)
  Outcome of HAE attacks for treatment with Cinryze (C1 inhibitor [human]) which was initiated more than 4 hours after onset of the attack will be reported.

SECONDARY OUTCOMES:
Time to Treatment For Attack | From enrollment through study participation (Approximately 13 years)
  Time to treatment for attack will be assessed. It is defined as the time between the onset of the attack and the first injection of treatment.
Time to Complete Resolution of Attack | From enrollment through study participation (Approximately 13 years)
  Time to complete resolution of attack will be assessed. It is defined as the time between the first injection of treatment and the complete resolution of all symptoms.
Total Duration of Attack | From enrollment through study participation (Approximately 13 years)
  Total duration of attack will be assessed. It is defined as the time between the onset of the attack and the complete resolution of all symptoms
Hereditary Angioedema-Treated Attacks | From enrollment through study participation (Approximately 13 years)
  The frequency, severity, and affected sites of HAE-treated attacks will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda Development Center Americas
Locations (74):
- Australia (2):
  - Campbelltown Hospital, Campbelltown, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
- Medizinische Universität Graz, Graz, Austria
- Faculdade de Medicina Do ABC, Santo André, São Paulo, Brazil
- Fakultni nemocnice u sv. Anny v Brne, Brno, Czechia
- Odense Universitetshospital, Odense, Denmark
- France (20):
  - Hopital de Hautepierre, Strasbourg, Bas-Rhin
  - Hopital Cote de Nacre, Caen, Calvados
  - Hopital Purpan, Toulouse, Haute-Garonne
  - CHU Angers, Angers
  - Centre Hospitalier Universitaire de Bordeaux, Hopital Pellegrin, Bordeaux
  - CHU La Cavale Blanche, Brest
  - CHU de GRENOBLE, Grenoble
  - Centre Hospitalier Le Mans, Le Mans
  - CHRU Lille, Lille
  - Groupement Hospitalier Edouard Herriot, Lyon
  - CHU Montpellier - Hôpital St Eloi, Montpellier
  - CHU de Nancy-Hopital Brabois Adulte, Nancy
  - Hôtel Dieu - Nantes, Nantes
  - CHU de Nice Archet I, Nice
  - Centre Hospitalier Georges Renon, Niort
  - Hôtel Dieu de Paris Hospital, Paris
  - Hôpital Saint Antoine, Paris
  - Hopital Cochin, Paris
  - CHU de Reims, Reims
  - Centre Hospitalier Universitaire de Saint Etienne, Saint-Etienne
- Germany (8):
  - Hals-Nasen-Ohrenklinik und Poliklinik, München, Bavaria
  - Klinikum der Johann-Wolfgang Goethe-Universitat, Frankfurt am Main, Hesse
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz, Rhineland-Palatinate
  - Universitätsklinikum Carl Gustav Carus an der TU Dresden, Dresden, Saxony
  - Charité - Universitätsmedizin Berlin, Berlin
  - Hämophilie Zentrum Rhein Main GmbH, Mörfelden-Walldorf
  - Universitätsklinikum Ulm, Ulm
- Greece (2):
  - Navy Hospital of Athens, Athens, Attica
  - Papageorgiou General Hospital of Thessaloniki, Thessaloniki
- St James's Hospital, Dublin, Ireland
- Israel (4):
  - Bnai Zion Medical Center, Haifa
  - Rabin Medical Center - PPDS, Petah Tikva
  - Sheba Medical Center - PPDS, Ramat Gan
  - Tel Aviv Sourasky Medical Center PPDS, Tel Aviv
- Italy (7):
  - AO Ospedale Policlinico Consorziale Di Bari, Bari, Apulia
  - Azienda Ospedaliero Universitaria Consorziale Policlinico di Bari, Bari, Apulia
  - Azienda Ospedaliera Universitaria Federico II, Napoli, Campania
  - ASST Fatebenefratelli Sacco - Ospedale Luigi Sacco, Milan, Lombardy
  - Presidio Policlinico Di Monserrato, Monserrato, Sardinia
  - Universita degli Studi di Padova, Padua
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia-Cervello, Palermo
- Spain (14):
  - CHUS - H. Clinico U. de Santiago, Santiago de Compostela, A Coruña
  - Hospital de La Marina Baixa, Villajoyosa, Alicante
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Vall d'Hebrón - PPDS, Barcelona
  - Hospital Cruz Roja Española de Gijón, Gijón
  - Hospital Universitario de Jaen, Jaén
  - Hospital de Santa Maria, Lleida
  - Centro de Alta Resolución de Procesos Asistenciales (C.A.R.P.A.), Logroño
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario La Paz - PPDS, Madrid
  - Hospital Universitario Virgen del Rocio - PPDS, Seville
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
  - Complejo Hospitalario Universitario de Vigo, Vigo
- Länssjukhuset Ryhov, Jönköping, Sweden
- United Kingdom (11):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire
  - John Radcliffe Hospital, Oxford, Oxfordshire
  - Frimley Park Hospital, Frimley, Surrey
  - St James University Hospital, Leeds, York
  - Birmingham Heartlands Hospital, Birmingham
  - University Hospital of Wales - PPDS, Cardiff
  - The Royal London Hospital, London
  - Royal Free Hospital, London
  - Manchester Royal Infirmary - PPDS, Manchester
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Maurer M, Aberer W, Caballero T, Bouillet L, Grumach AS, Botha J, Andresen I, Longhurst HJ; IOS Study Group. The Icatibant Outcome Survey: 10 years of experience with icatibant for patients with hereditary angioedema. Clin Exp Allergy. 2022 Sep;52(9):1048-1058. doi: 10.1111/cea.14206. Epub 2022 Aug 7. PMID 35861129
- [Derived] Guilarte M, Sala-Cunill A, Baeza ML, Cabanas R, Hernandez MD, Ibanez E, de Larramendi CH, Lleonart R, Lobera T, Marques L, de San Pedro BS, Botha J, Andresen I, Caballero T; IOS Study Group. Hereditary angioedema due to C1 inhibitor deficiency: real-world experience from the Icatibant Outcome Survey in Spain. Allergy Asthma Clin Immunol. 2021 Dec 29;17(1):137. doi: 10.1186/s13223-021-00641-3. PMID 34965883
- [Derived] Longhurst HJ, Dempster J, Lorenzo L, Buckland M, Grigoriadou S, Symons C, Bethune C, Fabien V, Bangs C, Garcez T. Real-world outcomes in hereditary angioedema: first experience from the Icatibant Outcome Survey in the United Kingdom. Allergy Asthma Clin Immunol. 2018 Aug 6;14:28. doi: 10.1186/s13223-018-0253-x. eCollection 2018. PMID 30127805
- [Derived] Caballero T, Zanichelli A, Aberer W, Maurer M, Longhurst HJ, Bouillet L, Andresen I; IOS Study Group. Effectiveness of icatibant for treatment of hereditary angioedema attacks is not affected by body weight: findings from the Icatibant Outcome Survey, a cohort observational study. Clin Transl Allergy. 2018 Mar 23;8:11. doi: 10.1186/s13601-018-0195-x. eCollection 2018. PMID 29599966
- [Derived] Aberer W, Maurer M, Bouillet L, Zanichelli A, Caballero T, Longhurst HJ, Perrin A, Andresen I; IOS Study Group. Breakthrough attacks in patients with hereditary angioedema receiving long-term prophylaxis are responsive to icatibant: findings from the Icatibant Outcome Survey. Allergy Asthma Clin Immunol. 2017 Jul 5;13:31. doi: 10.1186/s13223-017-0203-z. eCollection 2017. PMID 28690642
- [Derived] Zanichelli A, Longhurst HJ, Maurer M, Bouillet L, Aberer W, Fabien V, Andresen I, Caballero T; IOS Study Group. Misdiagnosis trends in patients with hereditary angioedema from the real-world clinical setting. Ann Allergy Asthma Immunol. 2016 Oct;117(4):394-398. doi: 10.1016/j.anai.2016.08.014. PMID 27742086
- [Derived] Longhurst HJ, Aberer W, Bouillet L, Caballero T, Maurer M, Fabien V, Zanichelli A; IOS Study Group. The Icatibant Outcome Survey: treatment of laryngeal angioedema attacks. Eur J Emerg Med. 2016 Jun;23(3):224-7. doi: 10.1097/MEJ.0000000000000292. PMID 27116379
- [Derived] Longhurst HJ, Aberer W, Bouillet L, Caballero T, Fabien V, Zanichelli A, Maurer M; IOS Investigators. Analysis of characteristics associated with reinjection of icatibant: Results from the icatibant outcome survey. Allergy Asthma Proc. 2015 Sep-Oct;36(5):399-406. doi: 10.2500/aap.2015.36.3892. PMID 26314822
- [Derived] Hernandez Fernandez de Rojas D, Ibanez E, Longhurst H, Maurer M, Fabien V, Aberer W, Bouillet L, Zanichelli A, Caballero T; IOS Study Group. Treatment of HAE Attacks in the Icatibant Outcome Survey: An Analysis of Icatibant Self-Administration versus Administration by Health Care Professionals. Int Arch Allergy Immunol. 2015;167(1):21-8. doi: 10.1159/000430864. Epub 2015 Jun 25. PMID 26112099
- [Derived] Maurer M, Longhurst HJ, Fabien V, Li HH, Lumry WR. Treatment of hereditary angioedema with icatibant: efficacy in clinical trials versus effectiveness in the real-world setting. Allergy Asthma Proc. 2014 Sep-Oct;35(5):377-81. doi: 10.2500/aap.2014.35.3780. Epub 2014 Aug 6. PMID 25198193
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fcf4db2bf003ab4684f